CLINICAL TRIAL: NCT05051865
Title: A Prospective, Single-center Clinical Study to Explore the Efficacy and Safety of Camrelizumab Combined With SHR1020 in the Treatment of Advanced Melanoma
Brief Title: To Explore the Efficacy and Safety of Camrelizumab Combined With SHR1020 in the Treatment of Advanced Melanoma
Status: Unknown | Phase: Phase 2 | Type: Interventional
Last Known Status: Recruiting
Sponsor: Peking University Cancer Hospital & Institute (Other)
Responsible Party: Principal Investigator, Jun Guo, Clinical Professor, Peking University Cancer Hospital & Institute
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: MM-IIT-SHR1210-FMTN
Record Dates: First submitted 2021-09-15; First posted 2021-09-21 (Actual); Last update posted 2022-11-17 (Actual); Status verified 2022-11

CONDITIONS: Melanoma
MeSH Terms: conditions — Melanoma | interventions — camrelizumab; famitinib

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Camrelizumab Combined With SHR1020 (Experimental): Camrelizumab combined with SHR1020 for advanced melanoma.
  Interventions: Drug: camrelizumab; Drug: SHR1020

INTERVENTIONS:
Drug: camrelizumab — camrelizumab combined with SHR1020 for advanced melanoma
  Other Names: SHR1210
Drug: SHR1020 — camrelizumab combined with SHR1020 for advanced melanoma

SUMMARY:
This study is being conducted to explore the efficacy and safety of camrelizumab combined with SHR1020 in the treatment of advanced melanoma.

DETAILED DESCRIPTION:
This trial is a prospective, single-center, single-arm clinical research. Based on current experience, single agent immunotherapy has limited efficacy in advanced melanoma. SHR1020 is a multi-target tyrosine kinase inhibitor. This study is aiming to evaluate the efficacy and safety of camrelizumab combined with SHR1020 in patients with advanced melanoma. The safety and efficacy of this study will be assessed through ORR, DCR, PFS, OS and adverse effects as graded by CTCAE 5.0.

ELIGIBILITY:
Inclusion Criteria:

* Has unresectable Stage III or Stage IV melanoma per American Joint Committee on Cancer (AJCC) staging system version 8. At least one measurable lesion conforming to RECIST 1.1 criteria.
* The toxicity of prior treatment has recovered to ≤1 grade according to CTCAE 5.0 (excepted alopecia).
* ECOG score 0-1.
* The expected survival time is ≥ 12 weeks.
* Had normal swallowing function, without dysfunction of gastrointestinal absorption.
* Adequate organ and bone marrow function.
* Female patients of childbearing age must undergo a serum pregnancy test within 7 days before the commencement of the study and the results are negative, and are willing to use a medically approved high potency contraceptive method during the study period and within 12 months after the last administration of the study drug; For male patients whose partner is a female of childbearing age, they should be surgically sterilized or agree to use an effective method of contraception during the study period and for 12 months after administration of the last study.
* Willing to consent and signed the informed consent, and able comply with the planned visit, research treatment, laboratory examination and other test procedures.

Exclusion Criteria:

* Other malignant tumors occurred in the past 5 years, except for cured skin basal cell carcinoma, squamous cell carcinoma of skin, early stage prostate cancer and cervical carcinoma in situ.
* Has uveal melanoma.
* The patient has previously received anti-angiogenic drugs.
* The first study drug treatment was less than 4 weeks from the last chemotherapy or 5 half-lives from the last targeted therapy; less than 4 weeks from major surgery; less than7 days from immunosuppressive drug; less than 3 weeks from immunomodulatory; less than 4 weeks from live attenuated vaccine.
* Systemic antibiotic use for 7 days within 4 weeks prior to initial administration, or unexplained fever during screening/prior to initial administration.
* Received hematopoietic stimulating factors (eg: G-CSF, EPO) within 1 week prior to initial administration.
* Patients with central nervous system disease or brain metastases; patients who have received treatment, such as imaging confirmed stable has been maintained for at least 4 weeks, and have stopped systemic hormone therapy for more than 2 weeks, no clinical symptoms can be included.
* With active autoimmune disease or a history of autoimmune disease.
* With history of allogeneic organ transplantation or allogeneic hematopoietic stem cell transplantation.
* With immunodeficiency, eg HIV, HBV, HCV.
* Known to be allergic to the active ingredients or excipients in this study.
* Have a clear history of serious and uncontrolled other disease or mental disorders.
* Has a bleeding tendency or abnormal clotting function (INR>2.0, PT>16s).
* Other situations that the researcher considers inappropriate to participate in the research.

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 60 (Estimated)
Dates: Start 2021-10-09 (Actual); Primary Completion 2024-08-30 (Estimated); Study Completion 2024-08-30 (Estimated)

PRIMARY OUTCOMES:
ORR (Objective Response Rate) | From date of first dose until the date of first documented progression or date of death from any cause, whichever came first, assessed up to 12 months
  Containing the incidence of complete response (CR) and partial response (PR). Evaluated according to RECIST 1.1 criteria, patients received their first tumor imaging evaluation at 6 weeks after the treatment start, followed by imaging evaluation every 2 cycles.

SECONDARY OUTCOMES:
PFS (Progression-Free-Survival) | From date of treatment start until the date of progression or the date of death due to any caus, assessed up to 12 months
  From date of treatment start until the date of progression or the date of death due to any cause. Evaluated according to RECIST 1.1 criteria, patients received their first tumor imaging evaluation at 6 weeks after the treatment start, followed by imaging evaluation every 2 cycles.
DCR (Disease Control Rate) | From date of first dose until the date of first documented progression or date of death from any cause, whichever came first, assessed up to 12 months
  Containing the incidence of complete response (CR), partial response (PR) and stable disease (SD).Evaluated according to RECIST 1.1 criteria, patients received their first tumor imaging evaluation at 6 weeks after the treatment start, followed by imaging evaluation every 2 cycles.
OS (overall survival) | From date of treatment start until the date of death from any cause or censored at the last day that the patient is documented to be alive, whichever came first, assessed up to 24 months
  From date of treatment start to any cause death or last follow-up.
6mPFS | Up to 6 months
  6-month- Progression-Free-Survival rate. Evaluated according to RECIST 1.1 criteria, patients received their first tumor imaging evaluation at 6 weeks after the treatment start, followed by imaging evaluation every 2 cycles.
Adverse events (per CTCAE v5.0 criteria) | Up to 12months
  To evaluate the adverse events of patients with advanced melanoma after treated with camrelizumab plus SHR1020.

CONTACTS AND LOCATIONS:
Overall Officials: Jun Guo, MD, Principal Investigator — Peking University Cancer Hospital & Institute
Locations (1):
- Beijing Cancer Hospital, Beijing, Beijing Municipality, China